CLINICAL TRIAL: NCT06394037
Title: Active Surveillance for Patients with Limited Ground-glass Nodules in China: a Prospective Multi-center Single-arm Trial (ECTOP-1028)
Brief Title: Active Surveillance for Limited GGNs
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Other Study IDs: ECTOP-1028
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-09

CONDITIONS: Lung Ground-glass Opacities; Active Surveillance
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation: Active surveillance
  Interventions: Procedure: Active surveillance

INTERVENTIONS:
Procedure: Active surveillance — Conduct thoracic computed tomography scans every 12 months. If progression occurs, the treamtent approach would involve surgery.

SUMMARY:
This study is a single-arm, multi-center, phase III trial conducted under the Eastern Cooperative Thoracic Oncoloy Project (ECTOP) . The primary objective of the study is to assess the 5-year overall survival of patients with one or two ground-glass opacities by employing an active surveillance approach rather than immediate surgical resection.

DETAILED DESCRIPTION:
The trial aims to confirm the hypotheses that delaying surgery until GGO nodules exhibit progression or meet certain criteria offers a prognosis equivalent to those undergoing immediate surgical resection, potentially allowing many of these patients to avoid surgery altogether.

ELIGIBILITY:
Patients eligible for enrollment in the study are required to meet all the following criteria.

1. Demonstrates the following on thin-section computed tomography (TSCT) scan:

   1. Presence of one or two GGNs (bilateral lesions are permitted).
   2. All lesions have remained stable without regression or enlargement for at least 3 months.
   3. The dominant lesion (the lesion with the largest maximum tumor diameter) has a maximum tumor diameter ≥0.6cm and ≤2cm.
   4. CTR ≤0.25 in lesions.
   5. No lymph node with a diameter >1cm in the mediastinal view.
   6. Not adjacent to the pleura in dominant lesion and no sign of pleural retraction in any lesions.
2. Has not previously undergo any anti-tumor drug or radiation therapy for the lung lesions.
3. Aged 18-75 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Written informed consent.

Patients will be excluded if they meet any of the following criteria.

1. History of any prior malignancies within the past 5 years.
2. History of lung surgery.
3. History of interstitial pneumonia, pulmonary fibrosis or other severe pulmonary diseases.
4. Presence of severe or uncontrolled diseases that may possibly reduce the 10-year life expectancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients visiting the hospitals/medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2038-05-01 (Estimated); Study Completion 2038-05-01 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  The event is defined as the death due to any causes.

SECONDARY OUTCOMES:
10-year overall survival | 10 years
  The event is defined as the death due to any causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical data including patient characteristics, CT images and pathology images.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years from the study end.
Access Criteria: Medical oncologists and surgeons who are interested in the study. Emails could be sent to the address below to obtain the shared data:
  hqchen1@yahoo.com